CLINICAL TRIAL: NCT05021757
Title: New Enrollment Post Approval Registry for the Shockwave Intravascular Lithotripsy (IVL) System With Shockwave C2 Coronary Intravascular Lithotripsy (IVL) Catheter
Brief Title: Disrupt CAD III Post-Approval Study (PAS)
Status: Completed | Type: Observational
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 64647
Record Dates: First submitted 2021-08-03; First posted 2021-08-25 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Intravascular Lithotripsy; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Disrupt CAD III PAS Cohort: Patients in the CathPCI Registry who undergo a PCI procedure using a Shockwave C2 Coronary IVL catheter and meeting the eligibility criteria will be included in the PAS cohort.
  Interventions: Device: Shockwave C2 Coronary IVL

INTERVENTIONS:
Device: Shockwave C2 Coronary IVL — PCI procedure using a Shockwave C2 coronary IVL catheter

SUMMARY:
The study design is a prospective, multicenter, observational, single-arm post-approval study using data collected in the National Cardiovascular Data Registry (NCDR®) CathPCI Registry®.

DETAILED DESCRIPTION:
Subject Population: Patients ≥18 years of age with severely calcified, stenotic de novo coronary artery lesions presenting with stable, unstable, or silent ischemia that are suitable for percutaneous coronary intervention (PCI) and with clinical characteristics similar to the Disrupt CAD III IDE study. Approximately 1000 patients in the CathPCI Registry® (including a minimum of 30 patients with permanent pacemakers [PPM] or implantable cardioverter defibrillators [ICDs]) will be enrolled. Subjects will be followed through discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI
3. Left ventricular ejection fraction >25% within 6 months
4. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
5. LAD, RCA or LCX (or of their branches) with:

   * Stenosis of ≥70% and <100% or
   * Stenosis ≥50% and <99% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve (FFR) value ≤0.80, or iFR <0.90 or IVUS or OCT minimum lumen area ≤4.0 mm²
6. The lesion length must not exceed 40 mm
7. The target vessel must have TIMI flow 3 at baseline (visually assessed; may be assessed after pre-dilatation)
8. Evidence of calcification at the lesion site by angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location

Exclusion Criteria:

1. Subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure
2. New York Heart Association (NYHA) class III or IV heart failure
3. Renal failure with serum creatinine >2.5 mg/dL or chronic dialysis
4. Subjects in cardiogenic shock or with clinical evidence of acute heart failure
5. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
6. Previous stent within target lesion (in-stent restenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severely calcified, stenotic de novo coronary artery lesions presenting with stable, unstable, or silent ischemia that are suitable for percutaneous coronary intervention (PCI) and with clinical characteristics similar to the Disrupt CAD III IDE study.
Sampling Method: Non-Probability Sample
Enrollment: 1212 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- American College of Cardiology/National Cardiovascular Data Registry (NCDR), Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disrupt CAD III PAS Cohort
Started | 1212
Completed | 1212
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 1212
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330
  Male | 882
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data is Unknown or Not Reported for some patients because Race is an optional field in the CathPCI registry data collection form.
  Participants
    American Indian or Alaska Native | 2
    Asian | 36
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 68
    White | 1060
    More than one race | 2
    Unknown or Not Reported | 42
Region of Enrollment [Number; unit: participants]
  United States | 1212

OUTCOME MEASURES:

1. Primary Outcome: All-cause Death Rate
Time Frame: Up to hospital discharge, approximately 24-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 1212
Participants | 3

2. Primary Outcome: Number of Participants With Procedure-related Adverse Events
Time Frame: Up to hospital discharge, approximately 24-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 1212
Participants | 35

3. Primary Outcome: Number of Participants With IVL-related Ventricular Arrhythmia
Time Frame: Up to hospital discharge, approximately 24-48 hours
Population: Information on IVL-specific data points were collected on a separate optional IVL Auxiliary data collection form in the CathPCI Registry. There were 153 subjects in the PAS cohort with available IVL Auxiliary data.
Measure: Count of Participants; unit: Participants
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 153
Participants | 0

4. Primary Outcome: Number of Participants With IVL Balloon Loss of Pressure/Rupture
Time Frame: Up to hospital discharge, approximately 24-48 hours
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 153
Participants | 2

5. Primary Outcome: Number of Participants With Serious Coronary Dissection Following Balloon Loss of Pressure/Rupture
Time Frame: Up to hospital discharge, approximately 24-48 hours
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 153
Participants | 0

6. Primary Outcome: Number of IVL-related Pacing Issues in Patients With PPM/ICD
Description: Events that may indicate an adverse device interaction including inappropriate inhibition of pacing during IVL device utilization, inappropriate ICD shock during IVL device utilization (for ICD patients only), and the need for device re-programming associated with IVL use (during or post procedure).
Time Frame: Up to hospital discharge, approximately 24-48 hours
Population: Information on IVL-specific data points in PPM/ICD patients were collected on a separate optional IVL Auxiliary data collection form in the CathPCI Registry. There were 12 subjects with PPM/ICD devices in the PAS cohort with available IVL Auxiliary data.
Measure: Count of Participants; unit: Participants
Arm/Group | Disrupt CAD III PAS Cohort
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to hospital discharge, approximately 24-48 hours
Description: In the CathPCI registry data collection form, intra- and post-procedure adverse events are captured in a pre-specified list. Information on procedure and device-relatedness, as well as serious or non-serious designation, is not captured in the registry.
Groups:
- Disrupt CAD III PAS Cohort: Patients in the CathPCI Registry who undergo a PCI procedure using a Shockwave C2 Coronary IVL catheter and meeting the eligibility criteria will be included in the PAS cohort. A minimum of 150 patients with 30-day follow-up will be included in the PAS cohort.
  Shockwave C2 Coronary IVL: PCI procedure using a Shockwave C2 coronary IVL catheter
Arm/Group | Disrupt CAD III PAS Cohort
All-Cause Mortality (participants affected / at risk) | 3/1212
Serious Adverse Events (participants affected / at risk) | 35/1212
Other Adverse Events (participants affected / at risk) | 0/1212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disrupt CAD III PAS Cohort (N=1212)
Coronary Artery Perforation (Cardiac disorders) | 7 (7)
Significant Coronary Artery Dissection (C and above) (Cardiac disorders) | 5 (5)
Bleeding - Access Site (Injury, poisoning and procedural complications) | 2 (2)
Bleeding - Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Bleeding - Hematoma at Access Site (Injury, poisoning and procedural complications) | 3 (3)
Bleeding - Other (Injury, poisoning and procedural complications) | 1 (1)
Bleeding - Retroperitoneal (Injury, poisoning and procedural complications) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 6 (6)
Heart Failure (Cardiac disorders) | 5 (5)
Myocardial Infarction (Cardiac disorders) | 8 (8)
New Requirement for Dialysis (Renal and urinary disorders) | 2 (2)
Other Vascular Complications Requiring Treatment (Vascular disorders) | 6 (6)
Stroke - Ischemic (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT05021757/Prot_SAP_000.pdf